CLINICAL TRIAL: NCT06246292
Title: Erector Spinae Plane Block: Anatomical Landmark Versus Ultra-sounded Guided Technique, a Randomized Controlled Trial
Brief Title: The Efficacy and Safety of Landmark-guided Compared to Ultrasound-guided Erector Spinae Plane Block Techniques for Analgesia in Female Patients After Breast Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB number: 00012098
Record Dates: First submitted 2024-01-27; First posted 2024-02-07 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-01

CONDITIONS: Nerve Block
Keywords: Nerve block; breast surgery; analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- landmark guided ESPB technique (Experimental): The ESPB was performed using the landmarks described by Vadera et al. (5). Before initiating the block procedure, the spinous process of the T4 vertebra and a point situated 3 cm to its side are marked at the appropriate level. The needle was inserted perpendicularly to the skin and advanced in all planes until it contacts the vertebra's transverse process. The depth at which the thoracic vertebra's transverse process lies from the skin can vary, ranging from 2 to 4 cm, contingent upon the individual's physique. The needle tip was positioned between the erector spinae muscle and the transverse process. The volume of local anesthetics was injected in this plane.
  Interventions: Procedure: Anatomical landmark-guided ESPB
- ultrasound-guided ESPB technique (Active Comparator): The block was performed based on the original description by Forero et al. (2). A high-frequency linear transducer (MyLab 70 Xvision, Esaote SpA, Florence, Italy) was positioned in the parasagittal plane 2 cm lateral to the T4 vertebra. Once the transverse process and the overlying erector spinae muscle were visible on the ultrasound, the needle was introduced using the in-plane technique. The needle was inserted in the cranial-to-caudal direction until it reached the tip of the transverse process. Following a negative aspiration and a successful hydro dissection, the local anesthetic solution was injected beneath the erector spinae muscle's fascia.
  Interventions: Procedure: Ultrasound-guided ESPB

INTERVENTIONS:
Procedure: Ultrasound-guided ESPB — The ESPB is a truncal block guided by ultrasound, involving the injection of local anesthetic beneath the erector spinae muscle (ESM), positioned between the ESM and the transverse process (TP) of the vertebra.
  Arms: ultrasound-guided ESPB technique
Procedure: Anatomical landmark-guided ESPB — The ESPB is a truncal block guided by anatomical landmarks, involving the injection of local anesthetic beneath the erector spinae muscle (ESM), positioned between the ESM and the transverse process (TP) of the vertebra.
  Arms: landmark guided ESPB technique

SUMMARY:
The erector spinae plane (ESP) block is a technique that helps alleviate acute pain. It involves injecting local anesthetic between the erector spinae muscle (ESM) and the vertebra's transverse process (TP). This technique can be guided by ultrasound or anatomical landmarks, and it can be performed while the patient is lying down, sitting or on their side.

DETAILED DESCRIPTION:
Ultrasound guidance has established itself as the norm for regional anesthesia procedures, enabling live visualization of anatomical structures and enhancing the precision and safety of needle insertion. Conversely, the blind technique relies on anatomical landmarks and the ability to palpate to direct needle insertion. Although the blind technique might provide simplicity and efficiency, uncertainties persist concerning its precision and possible associated risks. As the popularity of the ESPB increases, a relevant query emerges: Should it be conducted with ultrasound guidance or through a non-guided technique? This study was designed to validate the efficacy and safety of a landmark-guided ESPB technique compared to an ultrasound-guided ESPB technique for analgesia in breast surgery. The hypothesis was that the ultrasound and anatomical landmark techniques for ESPB would provide equivalent analgesia. The study's primary objective was to compare the success rate of both techniques. The secondary objectives were to compare the dermatomal block spread, analgesic effectiveness, and technique-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Patients had an American Society of Anesthesiology (ASA) physical score of I-II.
* Patients undergoing unilateral elective breast surgery.

Exclusion Criteria:

* Patients had a contraindication to an ESPB (including coagulopathy, recent anticoagulant medication usage, or infection at the needle puncture site).
* Patients had a history of opioid addiction, preoperative opioid use, and allergies to study medications.
* Obesity (body mass index exceeding 35 kg/m²).
* If the placement of ESPB was not completed due to technique difficulties.
* Patients who expressed a lack of willingness to participate in the study were not considered eligible for participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
To compare the success rate of both landmark-guided ESPB and ultrasound-guided ESPB techniques for analgesia in breast surgery | 30 minutes after regional block procedure
  The primary outcome was the binary outcome: therapeutic success or failure of ESPB techniques in achieving cutaneous sensory block for breast surgery (from T1 to T6).

SECONDARY OUTCOMES:
To compare the dermatomal block spread in both groups | 30 minutes after regional block procedure.
  Assessment of the number of blocked cutaneous sensory dermatomes from T1 to T10.
To compare the analgesic effectiveness in both groups | The first 24 hours postoperatively at 1, 3, 6, 12, and 24 hours.
  Assessment of rest visual analog score (VAS) for surgical site pain (0 -10) 2.
To compare the technique-related complications in both groups | During the regional block procedure.
  Assessment of occurrence of adverse effects.
To compare the analgesic effectiveness in both groups | The first 24 hours postoperatively.
  The time (minutes) to the first intravenous patient-controlled analgesia (IV-PCA) demand dose.
To compare the analgesic effectiveness in both groups | intra- and 24 hours postoperatively
  Total fentanyl opioid consumption (microgram).

CONTACTS AND LOCATIONS:
Overall Officials: Islam elbardan, Dr., Principal Investigator — University of Alexandria
Locations (1):
- faculty of medicine, Alexandria Unverisity, Alexandria, Egypt